CLINICAL TRIAL: NCT05608915
Title: External vs Internal-triggered Augmented-reality Visual Cues to Treat Freezing of Gait
Acronym: ELIMINATE-FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Parkinson's Disease Association, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-846
Record Dates: First submitted 2022-10-31; First posted 2022-11-08 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic; Parkinsonian Disorders; Movement Disorders; Gait, Unsteady; Gait, Festinating
Keywords: Parkinson disease; Freezing of gait; FOG; PD; augmented reality; cue; cueing; visual; gait freezing
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Parkinsonian Disorders; Movement Disorders

STUDY DESIGN:
Intervention Model Description: All participants will receive all interventions in a crossover fashion, on the same day. All participants will first experience the conventional cue intervention. The order of the remaining interventions will be randomized. All conditions will be performed after participants hold (do not take) their morning dopaminergic medications.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented-Reality Visual Cues (Experimental): In this single-arm study, all participants will receive all interventions on the same day. They will be wearing an augmented-reality headset that will display a digital obstacle course. Walking performance will be captured with no visual cues, with conventional visual cues, and with augmented-reality visual cues.
  Interventions: Other: No Cue; Other: Conventional Cue; Other: Constant Cue; Other: Patient hand-triggered; Other: Patient eye-triggered; Other: Examiner-triggered

INTERVENTIONS:
Other: No Cue — There will be no visual cues at all. Will be tested off-medication (after holding morning dopaminergic medications).
Other: Conventional Cue — Physical lines taped to floor at regular intervals. Will be tested off-medication (after holding morning dopaminergic medications).
Other: Constant Cue — The augmented-reality visual cue will always be turned on. Will be tested off-medication (after holding morning dopaminergic medications).
Other: Patient hand-triggered — The augmented-reality visual cue will be turned on, intermittently, each time the patient clicks a handheld button. Will be tested off-medication (after holding morning dopaminergic medications).
Other: Patient eye-triggered — The augmented-reality visual cue will be turned on, intermittently, each time the patient looks down at the floor near their feet. Will be tested off-medication (after holding morning dopaminergic medications).
Other: Examiner-triggered — The augmented-reality visual cue will be turned on, intermittently, by an examiner, whenever they feel the patient is having a freezing episode or at risk of having a freezing episode. Will be tested off-medication (after holding morning dopaminergic medications).

SUMMARY:
Postural instability, freezing-of-gait (FOG), and falls are among the greatest unmet needs in Parkinson disease (PD). FOG eventually affects more than half of people with PD, and is notoriously difficult to treat pharmacologically or via deep brain stimulation. Visual cues do improve gait freezing, but their efficacy and adoption is limited because they are not practical to use in all real-world situations. There is a need for a cueing technique that is on-demand and discreet - only perceptible to the patient. Fortunately, recent technological advances in augmented-reality (AR) enable such an approach. In this study, state-of-the-art AR glasses will be used to project digital cues that are only visible to the wearer, to determine if they can improve FOG. 36 individuals with PD and FOG will be recruited to perform an obstacle-course gait task under six cue conditions: no cue, conventional cue, constant-on AR, patient-hand-triggered AR (turns on when patient clicks button), patient-eye-triggered AR (turns on when looking down), and examiner-triggered AR. The AR cue is a set of images that appear on the floor at a patient's feet, mimicking floor lines. Gait performance will be captured on video and via body-worn wireless sensors that detect how each limb is moving. The investigators will determine whether individuals are cue-able with conventional visual cues, whether intermittent cues outperform constant-on cues, and whether cues triggered by an examiner outperform cues triggered by patients themselves.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD
* Presence of freezing of gait, defined as a score of ≥1 in MDS-UPDRS 2.13, or 3.11.
* Can walk without assistance, OFF meds, based on yes/no verbal response

Exclusion Criteria:

* Severity of gait impairment should not require dependency to walker or cane
* Concomitant conditions that may affect significantly the evaluation of balance or gait, including orthopedic, rheumatologic or other neurological diseases
* Contraindication to physical therapy
* Severe bilateral visual impairment
* Age < 21
* Diagnosis of dementia
* Not agreeable to having video taken of entire research visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Stride Time Coefficient of Variation | For each arm, during the single-day research visit only.
  Marker of gait dysfunction, derived from kinematic recordings from body-worn wireless sensors.
Percent Time Freezing | For each arm, during the single-day research visit only.
  Marker of gait freezing, derived from video recordings of gait performance, and body-worn wireless sensors.

SECONDARY OUTCOMES:
Step Cadence | For each arm, during the single-day research visit only.
  Marker of dysfunction, derived from kinematic recordings from body-worn wireless sensors.
Gait Velocity | For each arm, during the single-day research visit only.
  Marker of gait dysfunction, derived from kinematic recordings from body-worn wireless sensors.
Mean Stride Length | For each arm, during the single-day research visit only.
  Marker of gait dysfunction, derived from kinematic recordings from body-worn wireless sensors.
Total Distance Walked | For each arm, during the single-day research visit only.
  Marker of gait dysfunction, derived from augmented-reality headset and other body-worn wireless sensors
Freezing Index | For each arm, during the single-day research visit only.
  Marker of gait freezing, derived from kinematic recordings from body-worn wireless sensors.
Number of Freeze Episodes | For each arm, during the single-day research visit only.
  Marker of gait freezing, derived from video recordings of gait performance, and body-worn wireless sensors.

CONTACTS AND LOCATIONS:
Overall Officials: James Liao, MD PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
At time of publication, a point of contact individual on the study team will be identified. Third parties will be able to request access to de-identified data used to support the publication findings by application to the Cleveland Clinic IRB. A data use agreement will be put in place between the CCF Cleveland Clinic and this third party for approved use of the data.